CLINICAL TRIAL: NCT02323685
Title: Single Escalating-dose, Open-label Study to Assess the Safety and Effect of SANGUINATE™ Infusion in Patients at Risk of Delayed Cerebral Ischemia (DCI) After Acute Aneurysmal Subarachnoid Hemorrhage (SAH)
Brief Title: Safety and Effect of SANGUINATE™ Infusion in Patients at Risk of Delayed Cerebral Ischemia (DCI) Following Subarachnoid Hemorrhage (SAH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: SGCI-002
Record Dates: First submitted 2014-11-12; First posted 2014-12-23 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Cerebral Ischemia
Keywords: DCI; Delayed Cerebral Ischemia; SAH; Subarachnoid Hemorrhage; Aneurysmal Subarachnoid Hemorrhage; Cerebral Ischemia; Brain Ischemia
MeSH Terms: conditions — Brain Ischemia; Subarachnoid Hemorrhage | interventions — PEGylated carboxyhemoglobin bovine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SANGUINATE™ (Experimental): Single infusion of SANGUINATE (pegylated carboxyhemogloblin)
  Interventions: Biological: SANGUINATE™

INTERVENTIONS:
Biological: SANGUINATE™ — Single infusion of SANGUINATE (pegylated carboxyhemogloblin)

SUMMARY:
Safety and effect of SANGUINATE on patients DCI following SAH.

DETAILED DESCRIPTION:
The purpose of this study is to study the safety and effect of SANGUINATE on patients suffering from delayed cerebral ischemia after acute aneurysmal subarachnoid hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent by the subject or his/her legally authorized representative;
* Modified Rankin (mRankin) score of 0 or 1 prior to the onset of subarachnoid hemorrhage;
* Ruptured aneurysm secured by endovascular coil embolization or surgical clipping (the Procedure), not more than 72 hours after the onset of subarachnoid hemorrhage; and
* Hunt and Hess (H&H) grade 3 or 4, or World Federation of Neurological Surgeons (WFNS) score 3 or 4 prior to the Procedure, and Modified Fisher (mFisher) grade 3 or 4, prior to the Procedure; or
* Clinical signs of ("symptomatic") delayed cerebral ischemia; or
* Angiographic evidence of cerebral vasospasm

Exclusion Criteria:

* In the judgment of the Investigator the patient is not a good candidate for the study
* Evidence of rebleed following the Procedure
* Subarachnoid hemorrhage secondary to trauma or to arteriovenous malformation
* Diagnosed moderate to severe pulmonary hypertension
* Radiologically confirmed moderate to severe pulmonary edema (as shown by the presence of Kerley lines, peribronchial cuffing, thickened interlobar fissure, consolidation and/or pleural effusion)
* History within the past 6 months and/or finding of decompensated heart failure
* Acute myocardial infarction within 3 months prior to the administration of the study drug
* Left ventricular ejection fraction <40%, as determined by prior echocardiography or clinical signs of CHF
* Medical history or concurrent evidence of moderate to severe renal insufficiency (estimated creatinine clearance < 30 mL/min)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-12; Primary Completion 2016-06 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Safety of study drug during and following infusion as measured by vital signs, clinical signs, bioanalytical measures, or investigational drug-related adverse events | Up to 30 days
  Safety assessments to include vital signs, clinical signs, bioanalytical measures, or investigational drug-related adverse events
Impact of SANGUINATE on brain oxygenation and blood flow assessed using Postitron Emission Tomography (PET) | Up to 30 days
  Blood oxygenation and blood flow will be assessed using Postitron Emission Tomography (PET)

SECONDARY OUTCOMES:
Changes in neurological function measured by National Institutes of Health Stroke Scale (NIHSS) | Up to 30 days
Incidence, location, and size of cerebral infarction as measured by MRI | Up to 30 days
Changes in Blood Gases as measured by Hemoximetry | Up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Michael N Dirringer, MD, Study Chair — Barnes Jewish Hospital/Washington University; Rajat Dhar, MD, Principal Investigator — Barnes Jewish Hospital/Washington University
Locations (1):
- Barnes Jewish Hospital/Washington University, St Louis, Missouri, United States